CLINICAL TRIAL: NCT01997229
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate the Safety and Efficacy of Eculizumab in Subjects With Refractory Generalized Myasthenia Gravis (gMG)
Brief Title: Safety and Efficacy of Eculizumab in Refractory Generalized Myasthenia Gravis (REGAIN Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ECU-MG-301; 2013-003589-15 (EudraCT Number)
Record Dates: First submitted 2013-11-18; First posted 2013-11-28 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Refractory Generalized Myasthenia Gravis
Keywords: Myasthenia Gravis; Eculizumab; safety; efficacy
MeSH Terms: conditions — Myasthenia Gravis | interventions — eculizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eculizumab (Experimental): Biological/Vaccine: Eculizumab; Induction phase: 3 vials of study drug (equivalent to 900 mg of eculizumab) weekly for 4 doses (every 7 days ± 2 days) followed by 4 vials of study drug (equivalent to 1200 mg of eculizumab) 1 week later for the fifth dose (Week 4); Maintenance phase: 4 vials of study drug (equivalent to 1200 mg of eculizumab) every 2 weeks (14 days ± 2 days) from the fifth dose onwards (Week 6 through Week 26).
  Interventions: Biological: Eculizumab
- Placebo (Placebo Comparator): Placebo contains the same buffer components without the active ingredient; Induction phase: 3 vials of study drug (placebo) weekly for 4 doses (every 7 days ± 2 days) followed by 4 vials of study drug (placebo) 1 week later for the fifth dose (Week 4); Maintenance phase: 4 vials of study drug (placebo) every 2 weeks (14 days ± 2 days) from the fifth dose onwards (Week 6 through Week 26).
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Eculizumab — Induction Phase: 900 mg IV weekly X 4 Maintenance Phase: 1200 mg IV every 2 weeks during Weeks 4-26
  Arms: Eculizumab
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if eculizumab is safe and effective for the treatment of refractory generalized Myasthenia Gravis.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female patients ≥18 years old
* Diagnosis of MG made by the following tests:

  1. Positive serologic test for anti-AChR Abs as confirmed at screening, and
  2. One of the following:

     1. History of abnormal neuromuscular transmission test demonstrated by single-fiber electromyography (SFEMG) or repetitive nerve stimulation, or
     2. History of positive anticholinesterase test, e.g. edrophonium chloride test, or
     3. Subject has demonstrated improvement in MG signs on oral cholinesterase inhibitors, as assessed by the treating physician.
* MGFA Clinical Classification Class II to IV at screening.
* MG-ADL total score must be ≥6 at screening and Randomization (Day 1).
* Subjects who have:

  1. Failed treatment with at least two immunosuppressive agents. Or,
  2. Failed treatment with at least one immunosuppressive agent and require chronic plasma exchange or IVIg

Key Exclusion Criteria:

* History of thymoma or other neoplasms of the thymus
* History of thymectomy within 12 months prior to screening
* MGFA Class I or MG crisis at screening (MGFA Class V)
* Use of rituximab within 6 months prior to screening
* Use of IVIg or PE within 4 weeks prior to Randomization (Day 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2013-12; Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (114):
- United States (41):
  - University of Alabama, Birmingham, Alabama
  - University of California San Francisco-Fresno, Fresno, California
  - University of Southern California, Los Angeles, California
  - University of California-Irvine, Orange, California
  - University of California Davis Health System, Sacramento, California
  - California Pacific Medical Center, San Francisco, California
  - Stanford University School of Medicine, Stanford, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - University of Florida Health Science Center, Jacksonville, Florida
  - University of Miami School of Medicine, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Georgia Regents University, Augusta, Georgia
  - Medical Associates of North Georgia, Canton, Georgia
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa College of Medicine, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University School Of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Lahey Clinic Inc., Burlington, Massachusetts
  - Wayne State University School of Medicine, Detroit, Michigan
  - Las Vegas Clinic, Las Vegas, Nevada
  - Buffalo General Hospital, Buffalo, New York
  - Hospital For Special Surgery/New York Presbyterian Hospital Cornell Campus, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Duke University Health System, Durham, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Wesley Neurology Clinic, Cordova, Tennessee
  - Vanderbilt Medical Center, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas
  - Methodist Neurological Institute, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Washington, Seattle, Washington
- Argentina (2):
  - Hospital Italiano, Ciudad Autonoma, Buenos Aires
  - Instituto de Investigaciones Neurologicas Raul Carrea, FLENI, Ciudad Autonoma, Buenos Aires
- Australia (2):
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Belgium (3):
  - UZ Antwerpen, Edegem
  - AZ Sint-Lucas - Campus Sint-Lucas, Ghent
  - UZ Leuven, Leuven
- Brazil (5):
  - Hospital Mãe de Deus, Porto Alegre, Rio Grande do Sul
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - HUCFF-UFRJ - Hospital Universitário Clementino Fraga Filho - Universidade Federal do Rio de Janeiro, Rio de Janeiro
  - UNIFESP - Universidade Federal de São Paulo, São Paulo
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Neurological Institute, Montreal, Quebec
- Czechia (3):
  - Vseobecna fakultni nemocnice v Praze, Prague, Prague
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Ostrava, Ostrava - Poruba
- Denmark (2):
  - Århus Universitetshospital, Aarhus C
  - Rigshospitalet, København Ø
- Finland (2):
  - Helsingin yliopistollinen keskussairaala, Helsinki
  - Neuro NEO Oy, Turku
- France (4):
  - CHU de Nice Hôpital Pasteur 2, Nice, Alpes Maritimes
  - Groupe Hospitalier Pellegrin - Hôpital Pellegrin, Bordeaux, Gironde
  - Hopital Roger Salengro - CHU Lille, Lille, Nord
  - Hopital Neurologique Pierre Wertheimer, Bron, Rhone
- Germany (2):
  - LMU-Campus Innenstadt, Munich, Bavaria
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
- Greece (2):
  - Navy Hospital of Athens, Athens
  - General Hospital of Thessaloniki "G. Papanikolaou", Thessaloniki
- Hungary (2):
  - Jahn Ferenc Del-Pesti Korhaz, Budapest
  - Szegedi Tud.Egyetem Szent-Gyorgyi Albert Klin. Közp., Szeged
- Italy (9):
  - Policlinico di Catania, Catania
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Ospedale San Camillo IRCCS, Padua
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Umberto I Pol. di Roma-Università di Roma La Sapienza, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Ospedaliera Sant'Andrea - Università di Roma La Sapienza, Roma
  - Ospedale Santa Chiara, Trento
- Japan (11):
  - Chiba University Hospital, Chiba, Chiba
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Hanamaki General Hospitals, Hanamaki-shi, Iwate
  - NHO Sendai Medical Center, Sendai, Miyagi
  - NHO Nagasaki Kawatana Medical Center, Kawatana, Nagasaki
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Kinki University Hospital, Osakasayama-shi, Osaka
  - Osaka University Hospital, Suita-shi, Osaka
  - Toho University Ohashi Medical Center, Meguro-ku, Tokyo-To
  - Yamaguchi University Hospital, Ube-shi, Yamaguchi
- Netherlands (3):
  - Academisch Medisch Centrum, Amsterdam
  - Leiden Universitair Medisch Centrum, Leiden
  - Maastricht University Medical Center, Maastricht
- South Korea (4):
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul Metropolitan Government Seoul National University, Seoul
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario La Paz, Madrid
- Sweden (2):
  - Sahlgrenska Sjukhuset, Gothenburg
  - Karolinska Universitetssjukhuset - Solna, Stockholm
- Turkey (Türkiye) (5):
  - Hacettepe University Medical Faculty, Ankara
  - Karadeniz Tecnical Uni. Med. Fac., Istanbul
  - Dokuz Eylul University Medicine Faculty, Izmir
  - Kocaeli University Medical Faculty, Kocaeli
  - Ondokuz Mayıs University of Medicine, Samsun
- United Kingdom (3):
  - The Walton Centre, Liverpool, Merseyside
  - Queen Elizabeth Hospital, Birmingham, West Midlands
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Howard JF Jr, Barohn RJ, Cutter GR, Freimer M, Juel VC, Mozaffar T, Mellion ML, Benatar MG, Farrugia ME, Wang JJ, Malhotra SS, Kissel JT; MG Study Group. A randomized, double-blind, placebo-controlled phase II study of eculizumab in patients with refractory generalized myasthenia gravis. Muscle Nerve. 2013 Jul;48(1):76-84. doi: 10.1002/mus.23839. Epub 2013 Apr 30. PMID 23512355
- [Result] Howard JF Jr, Utsugisawa K, Benatar M, Murai H, Barohn RJ, Illa I, Jacob S, Vissing J, Burns TM, Kissel JT, Muppidi S, Nowak RJ, O'Brien F, Wang JJ, Mantegazza R; REGAIN Study Group. Safety and efficacy of eculizumab in anti-acetylcholine receptor antibody-positive refractory generalised myasthenia gravis (REGAIN): a phase 3, randomised, double-blind, placebo-controlled, multicentre study. Lancet Neurol. 2017 Dec;16(12):976-986. doi: 10.1016/S1474-4422(17)30369-1. Epub 2017 Oct 20. PMID 29066163
- [Derived] Monteleone JPR, Gao X, Kleijn HJ, Bellanti F, Pelto R. Eculizumab Pharmacokinetics and Pharmacodynamics in Patients With Generalized Myasthenia Gravis. Front Neurol. 2021 Nov 2;12:696385. doi: 10.3389/fneur.2021.696385. eCollection 2021. PMID 34795626
- [Derived] Siddiqi ZA, Nowak RJ, Mozaffar T, O'Brien F, Yountz M, Patti F; REGAIN Study Group. Eculizumab in refractory generalized myasthenia gravis previously treated with rituximab: subgroup analysis of REGAIN and its extension study. Muscle Nerve. 2021 Dec;64(6):662-669. doi: 10.1002/mus.27422. Epub 2021 Oct 14. PMID 34590717
- [Derived] Nowak RJ, Muppidi S, Beydoun SR, O'Brien FL, Yountz M, Howard JF Jr. Concomitant Immunosuppressive Therapy Use in Eculizumab-Treated Adults With Generalized Myasthenia Gravis During the REGAIN Open-Label Extension Study. Front Neurol. 2020 Nov 24;11:556104. doi: 10.3389/fneur.2020.556104. eCollection 2020. PMID 33329303
- [Derived] Mantegazza R, Wolfe GI, Muppidi S, Wiendl H, Fujita KP, O'Brien FL, Booth HDE, Howard JF Jr; REGAIN Study Group. Post-intervention Status in Patients With Refractory Myasthenia Gravis Treated With Eculizumab During REGAIN and Its Open-Label Extension. Neurology. 2021 Jan 26;96(4):e610-e618. doi: 10.1212/WNL.0000000000011207. Epub 2020 Nov 23. PMID 33229455
- [Derived] Mantegazza R, O'Brien FL, Yountz M, Howard JF Jr; REGAIN study group. Consistent improvement with eculizumab across muscle groups in myasthenia gravis. Ann Clin Transl Neurol. 2020 Aug;7(8):1327-1339. doi: 10.1002/acn3.51121. Epub 2020 Jul 22. PMID 32700461
- [Derived] Jacob S, Murai H, Utsugisawa K, Nowak RJ, Wiendl H, Fujita KP, O'Brien F, Howard JF Jr. Response to eculizumab in patients with myasthenia gravis recently treated with chronic IVIg: a subgroup analysis of REGAIN and its open-label extension study. Ther Adv Neurol Disord. 2020 May 6;13:1756286420911784. doi: 10.1177/1756286420911784. eCollection 2020. PMID 32426038
- [Derived] Vissing J, Jacob S, Fujita KP, O'Brien F, Howard JF; REGAIN study group. 'Minimal symptom expression' in patients with acetylcholine receptor antibody-positive refractory generalized myasthenia gravis treated with eculizumab. J Neurol. 2020 Jul;267(7):1991-2001. doi: 10.1007/s00415-020-09770-y. Epub 2020 Mar 18. PMID 32189108
- [Derived] Andersen H, Mantegazza R, Wang JJ, O'Brien F, Patra K, Howard JF Jr; REGAIN Study Group. Eculizumab improves fatigue in refractory generalized myasthenia gravis. Qual Life Res. 2019 Aug;28(8):2247-2254. doi: 10.1007/s11136-019-02148-2. Epub 2019 Mar 23. PMID 30905021
- See also: Alexion Clinical Trials Webpage — http://www.alexionclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Eculizumab: Induction phase: 3 vials of study drug (equivalent to 900 mg of eculizumab) weekly for 4 doses (every 7 days ± 2 days) followed by 4 vials of study drug (equivalent to 1200 mg of eculizumab) 1 week later for the fifth dose (Week 4).
  Maintenance phase: 4 vials of study drug (equivalent to 1200 mg of eculizumab) every 2 weeks (14 days ± 2 days) from the fifth dose onwards (Week 6 through Week 26).
- Placebo: Induction phase: 3 vials of study drug (placebo) weekly for 4 doses (every 7 days ± 2 days) followed by 4 vials of study drug (placebo) 1 week later for the fifth dose (Week 4).
  Maintenance phase: 4 vials of study drug (placebo) every 2 weeks (14 days ± 2 days) from the fifth dose onwards (Week 6 through Week 26).
Period: Overall Study
Arm/Group | Eculizumab | Placebo
Started | 62 | 63
Completed | 57 | 61
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eculizumab | Placebo | Total
Number analyzed (Participants) | 62 | 63 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (15.66) | 46.9 (17.98) | 47.2 (16.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 41 | 82
  Male | 21 | 22 | 43

OUTCOME MEASURES:

1. Primary Outcome: Myasthenia Gravis Activities of Daily Living Profile (MG-ADL): Change From Baseline in MG-ADL Total Score at Week 26 by Worst-Rank Analysis of Covariance (ANCOVA)
Description: In the Worst-Rank analysis, the 125 total patients were ranked from best outcome (rank/score of 1) to worst outcome (rank/score of 125).
Time Frame: End of study (Week 26)
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Eculizumab | Placebo
Number analyzed (Participants) | 62 | 63
scores on a scale | 56.6 (4.53) | 68.3 (4.49)
Statistical Analysis 1: Comparison: Eculizumab vs Placebo; Test type: Superiority; p = 0.0698, ANCOVA; Mean Difference (Net) = -11.7, 95% CI 2-sided [-24.33 to 0.96]

ADVERSE EVENTS:
Time Frame: 26 weeks (Study Period) + 8 weeks (Follow-up Period for subjects who discontinued the Study Period or completed the Study Period but did not enroll in the ECU-MG-302 extension trial)
Arm/Group | Eculizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/63
Serious Adverse Events (participants affected / at risk) | 9/62 | 18/63
Other Adverse Events (participants affected / at risk) | 52/62 | 53/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=62) | Placebo (N=63)
Deep vein thrombosis (Vascular disorders) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 5 | 8
Myasthenia gravis crisis (Nervous system disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Varicella (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=62) | Placebo (N=63)
Contusion (Injury, poisoning and procedural complications) | 5 | 2
Dizziness (Nervous system disorders) | 5 | 5
Headache (Nervous system disorders) | 10 | 12
Myasthenia gravis (Nervous system disorders) | 1 | 5
Paraesthesia (Nervous system disorders) | 3 | 4
Chills (General disorders) | 1 | 4
Oedema peripheral (General disorders) | 4 | 2
Insomnia (Psychiatric disorders) | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 8 | 8
Nausea (Gastrointestinal disorders) | 8 | 9
Vomiting (Gastrointestinal disorders) | 3 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2
Nasopharyngitis (Infections and infestations) | 9 | 10
Oral herpes (Infections and infestations) | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 10 | 10
Urinary tract infection (Infections and infestations) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication rights are tied to the completion of the multi-center publication.